CLINICAL TRIAL: NCT06662981
Title: The Effect of Preoperative Information and Education in the Clinical Outcome of Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, SARA ELENI AMPRACHIM, RN, MSc, MSc, PhD (c), General Hospital of Attica "KAT", Athens, Greece, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11000
Record Dates: First submitted 2023-09-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2023-09

CONDITIONS: Total Hip Arthroplasty
Keywords: preoperative information; preoperative education; total hip arthroplasty
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- preoperative education (Experimental): The intervention will include oral and written education about the operation, nursing and active participation in self-care. The intervention will take place in 3 phases: One week before THA, one day before THA after patient admission and postoperatively, before patient discharge. After a rough description of the operation, the anatomy and functionality of the joint will be presented, underlining the necessity of the operation. Instructions for recognizing and managing potential complications will be given. Patients will be informed about the appropriate post-operative walking aids, walking style, sitting up techniques, standing-up techniques, lying down techniques and getting in and out of the car. There will be a demonstration of muscle strengthening exercises, isometric quadriceps and gluteal exercises, Patients will also be informed about the necessity of prophylactic postoperative antithrombotic and antibiotic treatment.
  Interventions: Behavioral: preoparative information and education
- no preoparative education (basic information) (No Intervention): Patients will receive the standard preoperative care, which will not include formalized education beyond routine consent.

INTERVENTIONS:
Behavioral: preoparative information and education — The intervention will include oral and written education about the operation, nursing and active participation in self-care. The intervention will take place in 3 phases: One week before THA, one day before THA after patient admission and postoperatively, before patient discharge. After a rough description of the operation, the anatomy and functionality of the joint will be presented, underlining the necessity of the operation. Instructions for recognizing and managing potential complications will be given. Patients will be informed about the appropriate post-operative walking aids, walking style, sitting up techniques, standing-up techniques, lying down techniques and getting in and out of the car. There will be a demonstration of muscle strengthening exercises, isometric quadriceps and gluteal exercises, Patients will also be informed about the necessity of prophylactic postoperative antithrombotic and antibiotic treatment.
  Arms: preoperative education

SUMMARY:
Preoperative patient information and education is an essential aspect of modern surgical care, particularly for patients undergoing total hip arthroplasty (THA). This prospective, randomized trial aims to assess the effects of structured preoperative education and information on clinical outcomes in patients undergoing THA.

DETAILED DESCRIPTION:
A total of 100 patients will be randomized into two groups: the intervention group (n = 50) receiving standardized preoperative information and education, and the control group (n = 50) receiving standard preoperative care without a formal educational component. Postoperative outcomes, including pain, functionality, mobility, length of hospital stay (LOS), health-related quality of life, anxiety and depression will be compared between the 2 groups.

ELIGIBILITY:
Exclusion criteria in the study will be patients:

* under 50 years old
* with reduced mental abilities
* with a presence of mental illness
* who have had previous hip surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Hip pain and functionality | 30 days postoperatively
  Assessed using modified Harris Hip Score (mHHS), validated in Greek, one day preoperatively and one month postoperatively
Length of Hospital Stay | 30 days postoperatively
  Duration of hospitalization, measured in days
Anxiety and Depression | 30 days postoperatively
  Assessed using the Hospital Anxiety and Depression Scale (HADS), validated in Greek, one day preoperatively, one day before discharge from hospital, and one month postoperatively
Health-related quality of life | 30 days postoperatively
  Assessed using EQ-5D-5L index and EQ-5D-5L visual analog scale (VAS), validated in Greek one day preoperatively, one day before discharge from hospital, and one month postoperatively

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Sara Eleni Amprachim, Athens, Athens
  - KAT Hospital, Kifissia, Attica

IPD SHARING:
Plan to Share IPD: No
Patient data will be processed by the primary investigator

REFERENCES:
- [Background] Amprachim SE, Vlamis J, Nikolaou VS, Pneumaticos SG. Role of Preoperative Information and Education of Patients Undergoing Total Hip Arthroplasty: A Narrative Review of the Literature. Cureus. 2024 Aug 3;16(8):e66094. doi: 10.7759/cureus.66094. eCollection 2024 Aug. PMID 39224727